CLINICAL TRIAL: NCT01634516
Title: An Investigation of the Effectiveness of the Mediterranean Diet in Pregnant Women at Risk of Developing Allergy in Their Infants: Pilot Randomised Controlled Trial
Brief Title: Effectiveness of Mediterranean Diet Intervention in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heriot-Watt University (Other)
Collaborators: University of Edinburgh (Other)
Responsible Party: Principal Investigator, Dean A. Sewell, Senior Lecturer in Human Physiology and Metabolism, Heriot-Watt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HWU113821/UoE; CZG/2/558 (Other Grant/Funding Number: CSO)
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Allergy
Keywords: Diet; Pregnant
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary support (Experimental): Face to face intervention plus subsequent telephone support
  Interventions: Behavioral: Dietary support
- No dietary support (Placebo Comparator): No face to face intervention plus subsequent telephone support
  Interventions: Behavioral: No dietary support

INTERVENTIONS:
Behavioral: Dietary support — Face to face intervention plus subsequent telephone support
  Arms: Dietary support
Behavioral: No dietary support — No face to face intervention or subsequent telephone support
  Arms: No dietary support

SUMMARY:
There has been an increase in asthma and allergic disease prevalence, especially in children. Given the high prevalence, and the associated high disease burden and costs, there is an urgent need to identify effective strategies for the primary prevention of asthma and allergy. A systematic review of the literature has found strong supportive epidemiological evidence of a protective role for the Mediterranean Diet (MD).

The investigators aim is to undertake a pilot trial in a sample of pregnant women to establish recruitment, retention, a measurable change to a dietary intervention encouraging greater adherence to a MD during pregnancy, and acceptability of the dietary advice and diet modifications.

This pilot study will be a 2-arm randomised controlled trial (RCT) in a sample population of around 50 Scottish pregnant women.

This work ultimately aims to contribute to improving health outcomes through seeking to reduce the incidence of asthma and allergic problems. This pilot trial will prove invaluable in informing the subsequent planned definitive parallel group RCT.

DETAILED DESCRIPTION:
Aims

The primary aims of this pilot trial are to investigate rates of maternal recruitment and retention, and adherence with a MD during the latter two trimesters of pregnancy (i.e. weeks 12 to 36). The secondary aims are to determine whether there is any subsequent measurable change in the Mediterranean Diet score and whether the dietary advice and diet modifications are acceptable.

Research questions

1. What are the recruitment and retention rates of pregnant mothers whose infants are at high risk of atopic disease?
2. Is the advice and dietary modification acceptable to participants?
3. To what extent are mothers able to adhere to a MD?
4. Can a MD score be increased in pregnancy?
5. Can a measurable change in a biomarker of oxidative stress be detected as a result of adherence to a MD?
6. Can any increases in MD be sustained during pregnancy?

Design

1. Trial design This is a two-arm pilot RCT. Trial participants will be recruited from 2-3 hospitals/community treatment centres in Scotland.
2. Participant recruitment

   Pregnant women aged 16 years and above will be sent a letter of invitation, information for participants, and a consent form for the trial with their dating scan appointment by the hospital. Interested participants will be invited to contact the researcher by text, phone or email to discuss the project and answer any questions they may have; they will then be screened for eligibility to take part in the trial.

   Eligibility of high risk women is defined as: those with one or more first degree blood relatives with atopic dermatitis (eczema), a food allergy, allergic rhinitis (hay fever) or asthma, using the question 'Do you, the mother, or the father or sibling of the baby have an allergic disease: eczema, a food allergy, hay fever or asthma?' Responses will be recorded on the screening questionnaire.

   The researcher will send to the participant a food frequency questionnaire for completion at home and a urine container with instructions to fill the container on the day of the scan and bring it, with the Consent form and the completed FFQ along with them to hand over to the researcher. The urine specimen will be used for the analysis of markers of oxidative stress, antioxidant activity and nitric oxide (NO) synthesis. The researcher will greet the participant in the waiting area of the clinic prior to their dating scan where their consent form, urine sample and FFQ will be collected. After their scan, consenting eligible participants will complete a baseline MD questionnaire.
3. Intervention

   The intervention is a 15 minute dietary advice session directed at increasing the MD score, with subsequent telephone support sessions throughout the pregnancy.

   Intervention arm

   Mothers randomised to the intervention arm will meet with the project researcher when visiting the hospital for their first dating scan. After the scan, participants will receive a 15 minute dietary advice session, encouraging the consumption of particular foods that are consistent with the MD, and the key messages will be supplemented through written/visual materials, and through regular supportive telephone calls. No energy restrictions will be suggested. A £10 supermarket voucher will be given to the participants.

   The first follow-up by the researcher will be by telephone 12 weeks post-baseline MD questionnaire to inform them they will receive the second MD questionnaire and reply envelope for completion and return. A further supermarket voucher to the value of £10 will be sent to the participant on receipt of the completed form.

   Two weeks prior to the 24 weeks post-baseline MD questionnaire the project researcher will contact participants by phone and arrange a home visit. When visited at home by the researcher, a third MD questionnaire and second FFQ will be completed and handed to the researcher and a urine sample will be obtained.

   Free and continuous telephone access to the researcher will be available throughout the study.

   Control arm

   Mothers randomised to the control arm will meet with the project researcher when visiting the hospital for their first dating scan. The participant will not receive the 15 minute dietary advice session. A £10 supermarket voucher will be given to the participants. The first follow-up by the researcher will be by telephone 12 weeks post-baseline MD questionnaire to inform them they will receive the second MD questionnaire and reply envelope for completion and return. A further supermarket voucher to the value of £10 will be sent to the participant on receipt of the completed form.

   Two weeks prior to the 24 weeks post-baseline MD questionnaire the project researcher will contact participants by phone and arrange a home visit. When visited at home by the researcher, a third MD questionnaire and second FFQ will be completed and handed to the researcher and a urine sample will be obtained.
4. Randomisation

   Allocation to the intervention or control arm will be via pre-randomised sealed envelopes, based on a predetermined random number allocation, restricted by recruitment site. This restricted randomisation will be carried out by an independent statistician.
5. Follow-up Participants will be enrolled for a total of ~7 months (i.e. from 12-36 weeks of pregnancy).

Outcome measures

* Recruitment rate (i.e. the proportion of those invited to take part compared with the number of consenting women)
* Retention rate (i.e. the proportion of those starting the study to those finishing)
* Change in MD score from baseline to 24 and 36 weeks of pregnancy
* Change in oxidative stress and whole-body NO production
* Acceptability of dietary advice and diet modifications

ELIGIBILITY:
Inclusion Criteria:

* Pregnant in first trimester
* Age 16 years and above
* One or more first degree blood relatives of the baby with atopic dermatitis(eczema), food allergy, allergic rhinitis (persistent or intermittent) or asthma
* Willing to give informed consent

Exclusion Criteria:

* Age <16 years
* No first degree blood relatives of the baby with atopic dermatitis (eczema), food allergy, allergic rhinitis (persistent or intermittent) or asthma
* Recent (within the last 3 months) or current involvement in a dietary or supplementation trial
* Unable to give informed consent

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Recruitment rate of pregnant mothers whose infants are at high risk of atopic disease. | 4 months

SECONDARY OUTCOMES:
Mediterranean Diet score in pregnancy | 12 and 24 weeks post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dean A. Sewell, PhD, Principal Investigator — Heriot-Watt University; Aziz Sheikh, MBBS, MD, Study Chair — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - Leith Community Treatment Centre, Edinburgh, Scotland
  - St John's Hospital, Livingston, Scotland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sewell DA, Hammersley VS, Devereux G, Robertson A, Stoddart A, Weir C, Worth A, Sheikh A. Investigating the effectiveness of the Mediterranean diet in pregnant women for the primary prevention of asthma and allergy in high-risk infants: protocol for a pilot randomised controlled trial. Trials. 2013 Jun 14;14:173. doi: 10.1186/1745-6215-14-173. PMID 23768094
- [Background] Sewell DA, Hammersley VS, Robertson A, Devereux G, Stoddart A, Weir CJ, Worth A, Sheikh A. A pilot randomised controlled trial investigating a Mediterranean diet intervention in pregnant women for the primary prevention of allergic diseases in infants. J Hum Nutr Diet. 2017 Oct;30(5):604-614. doi: 10.1111/jhn.12469. Epub 2017 Feb 16. PMID 28211106